CLINICAL TRIAL: NCT02426580
Title: Dietary Education Intervention With Wechat Model Will Impact on Dietary Protein Intake in Patient Treated With Peritoneal Dialysis
Brief Title: Dietary Education Intervention Impact on Dietary Protein Intake in PD
Acronym: DIPIPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Second Affiliated Hospital of Chongqing Medical University (Other)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Principal Investigator, Dr. R. Gong, Director, chief physician, The Second Affiliated Hospital of Chongqing Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Chengdu 3rd Hospital
Record Dates: First submitted 2015-04-22; First posted 2015-04-27 (Estimated); Results first posted 2019-06-17 (Actual); Last update posted 2019-07-10 (Actual); Status verified 2019-07

CONDITIONS: Dietary Modification

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention with wechat group (Experimental): The wechat model will provide information of protein, calcium, phosphorus and sodium intake, which were suggested by the current KDIGO/ KDOQI guideline.
  Interventions: Behavioral: wechat
- Controlled group (No Intervention): Only conventional education every 3 months during routing clinical visit

INTERVENTIONS:
Behavioral: wechat — The wechat model of dietary education every 1 month by cellphone
  Other Names: wechat model
  Arms: Intervention with wechat group

SUMMARY:
This study is a prospective randomized controlled pilot trial/(a combined prospective and retrospective study). The investigators will use wechat intervening dietary protein intake in patients treated with peritoneal dialysis.

DETAILED DESCRIPTION:
Malnutrition is highly prevalent in peritoneal dialysis (PD) patients, and protein malnutrition will adversely affect outcomes. The investigators develop a dietary education intervention for PD patients to improve fundamental food knowledge that will increase protein intake to target level of 1.2 g/kg of protein intake per day. In additional the dietary intervention will provide information about sodium, phosphorus, calcium intake. To more effectively deliver the intervention, the investigators explored a technology using social media in China called wechat. The purpose of this study is to test whether a dietary intervention can be more effective when delivered using wechat compared to a traditional patient education intervention delivered during routing clinical visits.

ELIGIBILITY:
Inclusion Criteria:

* 1. All patients followed at the PD center who successful completed training and have received treatment for at least 1 month.
* 2. The life expectancy will be more than one year.
* 3. All patients will provide written informed consent.

Exclusion Criteria:

* 1.the patients will be severe ill status and unlikely to survive for 12 months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2018-05 (Actual)

IPD SHARING:
Plan to Share IPD: Yes
We would like to share the study protocol, study reports and informed consent form with other researchers.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: The data will become available at May 2019 and for 2 years
Access Criteria: No criteria.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were retrospectively from January 2014 to January 2015 and prospectively enrolled from Apr. 2015 to Apr. 2017 in the control group.
  Patients were prospectively enrolled in intervention with wechat group from Apr. 2015 to Apr. 2017.
Groups:
- Intervention With Wechat Group: The wechat model will provide information of protein, calcium, phosphorus and protein intake, which were suggested by the current KDIGO/ KDOQI guideline.
  wechat: The wechat model of dietary education every 1 month by cellphone
Period: Overall Study
Arm/Group | Intervention With Wechat Group | Controlled Group
Started | 70 (April 2015) | 70 (January 2014)
Completed | 59 (the last patient enrolled in this group in April 2017) | 54 (the last patient in this group enrolled in April 2017)
Not Completed | 11 | 16
Not completed — Death | 2 | 2
Not completed — Lost to Follow-up | 0 | 9
Not completed — transfer to hemodialysis | 5 | 5
Not completed — Kidney transplant | 3 | 0
Not completed — Allergic to egg white | 1 | 0

BASELINE CHARACTERISTICS:
Population: 11 (11/70, 15.71%) dropped out from intervention group and 16 (16/70, 22.86%) dropped out from control group; the rest of participants finished the study.
Groups:
- Controlled Group: Only conventional education every 3 months during routing clinical visit. The patients is Prospectively and retrospectively enrolled
- Total: Total of all reporting groups
Arm/Group | Intervention With Wechat Group | Controlled Group | Total
Number analyzed (Participants) | 59 | 54 | 113
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 59 | 54 | 113
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.3390 (13.8621) | 48.0926 (13.3985) | 47.17699 (13.61015)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 20 | 45
  Male | 34 | 34 | 68
Race (NIH/OMB) [Count of Participants; unit: Participants] — inquire of patients about race
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 59 | 54 | 113
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 0 | 0 | 0
    White | 0 | 0 | 0
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  China | 59 | 54 | 113
Normalized Protein Catabolic Rate (nPCR) [Mean (Standard Deviation); unit: g/(Kg*d)] — We use software (PD ADEQUEST 2.0) to conduct the Peritoneal Equilibration Test (PET) test. The result of PET test can offered the value of nPCR. nPCR can estimate daily protein intake of patients. Its units is g / (kg*d).
  g/(Kg*d) | 0.889 (0.202) | 0.862 (0.186) | 0.876 (0.194)

OUTCOME MEASURES:

1. Primary Outcome: Normalized Protein Catabolic Rate (nPCR)
Description: We use software (PD ADEQUEST 2.0) to conduct the Peritoneal Equilibration Test (PET) test. The result of PET test can offered the value of nPCR. nPCR can estimate daily protein intake of patients. Its units is g/(kg*d).
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: g/(kg*d)
Arm/Group | Intervention With Wechat Group | Controlled Group
Number analyzed (Participants) | 59 | 54
g/(kg*d) | 1.038 (0.188) | 0.930 (0.175)

ADVERSE EVENTS:
Time Frame: 1 year
Description: During the observation period of one year, all the enrolled participants were followed up per 1 to 3 months. And we recorded their disease status such as hospitalization, peritonitis, abdominal pain, rash and death.
Arm/Group | Intervention With Wechat Group | Controlled Group
All-Cause Mortality (participants affected / at risk) | 2/70 | 2/70
Serious Adverse Events (participants affected / at risk) | 0/70 | 0/70
Other Adverse Events (participants affected / at risk) | 1/70 | 0/70
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention With Wechat Group (N=70) | Controlled Group (N=70)
Egg white allergy (Gastrointestinal disorders) | 1 (1) | 0 (0) — In the intervention with wechat group, Only 1 patient had abdominal pain after eating egg white. And we considered this symptom caused by egg white allergy. Therefore, this patient excluded from the study

LIMITATIONS AND CAVEATS:
It is not a randomized controlled study. The patients assigned to both groups according to their willing. Most enrolled to intervention group. To improve the amount of control group, we retrospectively recruited 35 patients from recent 1 year.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-04-30): https://cdn.clinicaltrials.gov/large-docs/80/NCT02426580/Prot_SAP_000.pdf